CLINICAL TRIAL: NCT02019199
Title: Magnetic Resonance Imaging ( MRI) for Radiation Therapy Treatment Planning Evaluation of Lung, Liver and Pancreatic Motion.
Brief Title: Magnetic Resonance Imaging (MRI) in Motion
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00032595
Record Dates: First submitted 2013-12-18; First posted 2013-12-24 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Liver Cancer, Lung Cancer, Pancreatic Cancer
MeSH Terms: conditions — Liver Neoplasms; Lung Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is a research initiative established to explore the use of magnetic resonance imaging (MRI) as a tool for detecting organ motion as it pertains to planning radiation therapy.

DETAILED DESCRIPTION:
The goal with radiation therapy is to treat the defined tumor and spare the surrounding normal tissue from receiving dose above specified tolerance doses. There is evidence of improved local control and survival with higher doses of radiation, however, at the same time there is the need to spare normal tissues from higher doses of radiation. Technologies that allow the delivery of an increased radiation dose to the tumor while sparing normal tissue have the potential of improving the therapeutic ratio. However, the development of these technologies has been hampered by organ respiratory motion particularly in the case of the lungs and liver. Inadequate radiation coverage of a tumor secondary to organ motion can lead to delivering a lower dose to a portion of the tumor. Making the field of radiation larger to account for organ motion results in unnecessary radiation dose to surrounding healthy tissues. It is therefore desirable to document the extent of motion of the organ in question prior to carrying out the radiation treatment planning. The organ motion impacts directly on the radiation dose distribution in the treatment volume.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 21
* Patients with primary or metastatic tumors in the lungs, liver, or pancreas
* Patients undergoing a planning CT scan in the Department of Radiation Oncology with tumor motion assessment - planning 4D-CT ordered by the treating Radiation Oncologist
* Signed, specific informed consent prior to study entry

Exclusion Criteria:

* Any condition for which a MRI procedure is contraindicated including presence of metallic material in the body, such as pacemakers, non- MRI compatible surgical clips, shrapnel, etc
* Pregnant or breast-feeding women
* Subjects who have difficulty lying flat on their back for extended periods of time

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults males or females with primary or secondary cancer tumors of the lung, liver or pancreas
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2011-11; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the accuracy, robustness, and efficacy of MRI for tumor motion measurement. | During MRI approx 1 hour
  MRI and CT ( all subjects will have a standard of care CT scan) data in DICOM format will be collected for analysis using commercial or customized - developed software. Image quality will be assessed based on signal-to-noise (SNR), contrast-to-noise ratio (CNR), and the presence of image artifacts. Data to be computed include, but are not limited to, tumor volumes (gross tumor volume, internal target volume, planning target volume, etc.), tumor motion parameters (range, trajectory, frequency, variation, probability distribution, etc.), and treatment plan parameters (target coverage, dose-volume-histogram, etc.).
Tumor volume | During MRI approx 1 hour
  Free breathing/breath-hold MRI will be compared to free breathing/breath-hold CT
Tumor contrast-to-noise ratio (CNR) | During MRI approx 1 hour
  Difference between CNR is measured by 4D-MRI and 4D-CT
Tumor Motion | During MRI approx 1 hour
  Difference between tumor motion as measured by 2D cine-MRI vs 4D-MRI vs 4D-CT

CONTACTS AND LOCATIONS:
Overall Officials: Brian Czito, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States